CLINICAL TRIAL: NCT01397149
Title: A Phase I/II, Multi-centre Trial to Assess the Safety, Efficacy, and Pharmacokinetics of Eltrombopag, Administered to Thrombocytopenic Chronic Lymphocytic Leukemia Patients Prior to Alkylating Agents and/or Purine Analogue-based Therapy
Brief Title: Eltrombopag in Thrombocytopenic Chronic Lymphocytic Leukemia (CLL) Patients (CLL2S Study of GCLLSG)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of Ulm (Other)
Collaborators: GlaxoSmithKline (Industry); German CLL Study Group (Other); WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Responsible Party: Principal Investigator, Stephan Stilgenbauer, Prof. Dr. med., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLL2S; 2010-023022-20 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2011-07-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Lymphocytic Leukemia; Thrombocytopenia
Keywords: Chronic lymphocytic leukemia; Thrombocytopenia; Alkylating agents; Purine derivatives; TPO receptor agonist
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eltrombopag (Experimental): In phase II, patients will be randomized (2:1 eltrombopag : placebo) to receive either eltrombopag or placebo to explore the efficacy and confirm the safety of the identified eltrombopag dose from Phase I.
  Interventions: Drug: Eltrombopag
- Film coated tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Dosage form, frequency and duration exactly as experimental arm.
  Arms: Film coated tablet
Drug: Eltrombopag — Phase I:
  Single arm dose-escalation trial part, to test 4 doses of eltrombopag (75mg, 150mg, 225mg, 300mg) to find the appropriate, feasible dose to achieve a durable increase in platelet count (≥100,000/µl). Eltrombopag will be administered once daily at the respective dose level for 2 weeks (unless platelet counts rise to > 400,000/µl).
  Phase II:
  Patients will be randomized (2:1 eltrombopag : placebo) to explore the efficacy and confirm the safety of the identified dose level from Phase I. Eltrombopag/placebo will be administered before starting each cycle (and possibly following chemotherapy treatment depending on data from phase I), and will continue during all cycles of treatment until subjects finish chemotherapy (alkylating agents and/or purine analogue-based therapy). The schedule and days of eltrombopag dosing in Phase II will be determined based on data analyzed from Phase I.
  Other Names: Revolade; Promacta
  Arms: Eltrombopag

SUMMARY:
The aim of this study is to find the appropriate dose of eltrombopag in thrombocytopenic CLL patients, that shortens the duration of the thrombocytopenia and achieves platelet count of ≥ 100/nl prior to the start of chemotherapy containing alkylating agents and/or Purine Analogues.

DETAILED DESCRIPTION:
The study is divided in a Phase I and a Phase II part. The phase I part uses an open-label, dose escalation design in order to find the appropriate, feasible dose of eltrombopag to achieve a durable increase in platelet count.

In phase II, patients will be randomized (2:1 eltrombopag : placebo) to explore the efficacy and confirm the safety of the identified eltrombopag dose from Phase I. Eltrombopag/placebo will be administered before starting each cycle and will continue during all cycles of treatment until subjects finish treatment with chemotherapy. The schedule and days of eltrombopag dosing in Phase II will be determined based on data analyzed from Phase I, but will not exceed the defined maximum tolerable dose (MTD).

Severe thrombocytopenia is a frequently associated hematologic condition in patients with CLL. In the earlier stages of the disease, mild thrombocytopenia is common in approximately 25% of CLL patients. Later in the disease, the bone marrow will become more extensively infiltrated by the neoplastic cells, which results in more severe thrombocytopenia. Thrombocytopenia in patients with CLL could result from the disease, a packed marrow or from autoimmunity/ITP. For patients with CLL who develop severe thrombocytopenia, treatment options are limited and administration of platelet transfusions is common. Additionally, treatment of CLL patients with chemotherapy to treat the disease can be hampered due to severe thrombocytopenia. The clinical consequences of severe thrombocytopenia include an increased tendency for bleeding, probably due to thrombocytopenia, compromised hemostasis, and delayed administration of chemotherapy with the consequence of less optimal disease control.

Eltrombopag is an orally bioavailable small molecule TPO receptor (TPO-R) agonist being developed by GlaxoSmithKline (GSK) as a treatment for thrombocytopenia. Eltrombopag has been shown to stimulate platelet production and elevates platelet counts in healthy volunteers and in patients with chronic ITP, and in patients with thrombocytopenia related to hepatitis C virus (HCV) (Jenkins, Blood 2007; Bussel, NEJM 2007; McHutchinson NEJM 2007).

The optimal dose of eltrombopag for thrombocytopenic patients with CLL is currently unknown. As such, one objective of this study is to define a safe and effective dose of eltrombopag for thrombocytopenic patients with CLL prior to alkylating agent and/or fludarabine-based therapy. The eltrombopag doses proposed for administration in this study are 75 mg up to 300 mg once daily.

As a prerequisite for the trial, detailed studies have been performed in laboratory of the principal investigator on the in-vitro effects of eltrombopag on CLL cells regarding cell survival, differentiation and proliferation. The results suggest that eltrombopag is unlikely to act as a growth factor in CLL. Therefore clinical trials investigating its effect on platelet counts in CLL are warranted (Zenz T. et al., ASH 2009).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL (based immunophenotyping performed at the central reference laboratory of the GCLLSG in Cologne)
* Platelet count <50 000/μl at time of screening (measured and confirmed twice)
* Patient is planned to receive alkylating agents and/or fludarabine-based therapy as 2nd or higher-line treatment
* ECOG Performance Status of 0-2
* Age >= 18 years
* Signed written informed consent, according to ICH-GCP, and national/local regulation, prior to performing any study-specific procedures
* Negative pregnancy test and willingness to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* Able to understand and comply with protocol requirements and instructions and intend to complete the study as planned.
* Adequate renal function (creatinine must not exceed the upper limit of normal (ULN) reference range by more than 50%) at study entry
* Adequate liver function: bilirubin £ 1.5 times the upper limit of normal. ALT or AST <= 3 times the upper limit of normal without liver involvement with CLL and <= 5 times the upper limit of normal in case of the liver involvement with CLL
* Prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) must be within 80 to 120% of the normal range with no history of hypercoagulable state
* Total albumin must not be below the lower limit of normal (LLN) by more than 20%.

Exclusion Criteria:

* Thrombocytopenia that is primarily caused by ITP
* Refractory CLL: defined as treatment failure (failure to achieve a CR or PR) or disease progression within 6 months of last fludarabine and/or bendamustine based therapy. NOTE: Subjects refractory to rituximab monotherapy as last therapy are permitted
* No prior therapy for CLL
* Active autoimmune hemolytic anemia (AIHA) requiring corticosteroid therapy >100mg equivalent to hydrocortisone, or chemotherapy
* Platelet count > 50 000/μl at screening
* Richter's transformation
* CNS involvement of B-CLL
* Active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment
* Past or current malignancy other than CLL (with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix or breast) unless tumor was successfully treated with curative intent at least 2 years prior to trial entry
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months, congestive heart failure, etc.
* History of significant cerebrovascular disease
* Recurring venous thrombosis or pulmonary embolism
* Glucocorticoids unless given in doses <= 100 mg/day hydrocortisone (or equivalent dose of other glucocorticoids) and for exacerbations other than CLL (e.g. asthma)
* Known HIV positivity
* Active hepatitis B, C
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of eltrombopag.
* Subjects known or suspected of not being able to comply with a study protocol
* Patients with recent history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism) within the preceding 6 months. Patients with recurrent arterial or venous thromboembolic events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in platelet count | up to 7 months
  Time points of assessment:
  1 wk before treatment; 2-3 times/wk during treatment; 30d after end of treatment
  Treatment duration:
  * Phase I: Two weeks
  * Phase II: Eltrombopag is given as concomitant treatment to chemotherapy, with a max. duration of max. 6 cycles of 28 days each. The exact schedule of Eltrombopag administration will be determined after evaluation of Phase I results.

SECONDARY OUTCOMES:
Adverse events | up to 8 months
  Time points of assessment: 1 wk before and continously during treatment up to day 60 after last eltrombopag/placebo administration.
  Treatment duration: see primary outcome measure.
Change in vital signs | up to 7 months
  Time points of assessment: 1 wk before treatment; at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration. Treatment duration: see primary outcome measure.
Change in clinical laboratory parameters | up to 7 months
  Time points of assessment: 1 wk before treatment; at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration. Treatment duration: see primary outcome measure.
Bleeding events | up to 7 months
  Time points of assessment: 1 wk before treatment; at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration.
  Assessed by WHO bleeding scale. Treatment duration: see primary outcome measure.
Number of required platelet transfusions | up to 7 months
  Time points of assessment: 1 wk before treatment; at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration Treatment duration: see primary outcome measure.
Number of chemotherapy dose delay/dose reduction | up to 7 months
  Time points of assessment: 1 wk before treatment; at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration. In phase II only.
CLL overall response rate | up to 7 months
  Time points of assessment: at start of each chemotherapy cycle (Phase II); up to day 30 after last eltrombopag/placebo administration. In phase II only.
Time to CLL progression | up to 2 years
  In phase II only.
  Pre-defined subgroups based on the following stratification factors:
  * prior lines of treatment (1 vs. 2 vs. 3)
  * platelet count at baseline ≤ 30,000/µL vs > 30,000
Trough-level pharmacokinetics of eltrombopag | up to 6 months
  Assessment at day 1 of each week with eltrombopag administration.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Stilgenbauer, Prof. Dr., Principal Investigator — Universitätsklinikum Ulm, Medizinische Klinik III
Locations (10):
- Medizinische Universität Wien, Innere Medizin I, Abt. Hämatologie und Hämastaseologie, Vienna, Austria
- Germany (9):
  - Universitätsklinikum Köln; Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Carl Gustav Carus Med. Klinik und Poliklinik I, Dresden
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie und Internistische Onkologie, Erlangen
  - Universitätsklinikum; Klinik für Hämatologie, Essen
  - Klinikum Frankfurt (Oder) Medizinische Klinik I, Frankfurt (Oder)
  - Universitätsklinikum Schleswig-Holstein, II. Medizinische Klinik und Poliklinik im Städtischen Krankenhaus, Kiel
  - Onkologische Schwerpunktpraxis Leer-Emden, Leer
  - Städtisches Klinikum München GmbH, Klinikum Schwabing, Klinik für Hämatologie, Immunologie, Palliativmedizin, Infektiologie und Tropenmedizin, München
  - Universitätsklinikum Ulm, Medizinische Klinik III, Ulm